CLINICAL TRIAL: NCT05030792
Title: An Attention-Restorative Therapy (ART)-Based Virtual Reality Intervention to Address Cancer-Related Cognitive Impairments Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2021.056; HUM00199671 (Other: University of Michigan)
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer Survivorship; Cancer-related Cognitive Impairment
Keywords: Virtual reality; Breast Cancer Survivor; Attention Restorative Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ART VR 3 times/week (Experimental): ART VR practice for 30 minutes, at home, 3 times per week
  Interventions: Other: Attention-restorative therapy (ART)-based virtual reality (VR)
- ART VR 4 times/week (Experimental): ART VR practice for 30 minutes, at home, 4 times per week
  Interventions: Other: Attention-restorative therapy (ART)-based virtual reality (VR)

INTERVENTIONS:
Other: Attention-restorative therapy (ART)-based virtual reality (VR) — The ART-based VR intervention will be provided using an Oculus Go™ which is a commercially available, all-in-one VR headset with a handheld controller.

SUMMARY:
This study is to assess the feasibility of using a Virtual Reality (VR) headset to provide nature-based Attention-Restorative Therapy (ART) as treatment for cognitive impairment in post-treatment cancer survivors. At ART's foundation is the belief that exposure to nature can improve attention by fully engaging a person in a safe and relaxing experience. This intervention uses a VR headset to expose the participant to nature while overcoming some potential barriers of nature-based interventions like access, physical ability, and bad weather. The goal of this study is to understand if people are willing to use the VR headsets to experience nature virtually, if they find it helpful with cancer-related cognitive impairments (CRCI) symptoms and if they are satisfied with using it. Participants will be asked to use self-management materials (weekly home practice logs, Oculus Go™ and online questionnaires) for 6 weeks. Investigators hope to use information from this small feasibility study to study the effectiveness of the intervention in a larger group of cancer survivors and ultimately to help cancer survivors struggling with cognitive impairments.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥18
* Stage I-III breast cancer
* Reports a negative change in cognitive function since their cancer diagnosis and rate their cognitive fatigue using a single item questions as a ≥4 on a numeric rating scale of 0-10 for 1 month or more.
* Completed primary treatment (chemotherapy, radiation and/or surgery) ≥ 3 months but no more than 10 years prior to registration.
* May use concurrent adjuvant endocrine therapy and/or HER2-targeted therapy while on study.
* Ability to provide informed written consent.
* Ability to read and write English.
* Ability to be independent in decision making. Must respond No to "Do you have a guardian or blanket power of attorney for legal transactions?"

Exclusion Criteria:

* Other therapies intended to treat CRCI (allowed if person has been on them for 30 days prior to registration, and dose or treatment is not expected to change, and CRCI remains sufficiently uncontrolled per criteria of 4 or more on a 0 to 10 scale).
* Antidepressants (allowed if person has been on them for 30 days prior to registration, and dose or treatment is not expected to change, and CRCI remains sufficiently uncontrolled per inclusion criteria).
* Chronic oral or intravenous systemic steroid use (defined as being used on a regular basis or who have a problem that has required ongoing use of steroids in the last 180 days for greater than 7 days).
* Psychiatric disorder such as severe depression, bipolar disorder, obsessive compulsive disorder or schizophrenia. (Defined per medical history and/or patient self-report.)
* Pain requiring opioid pain medication.
* Electronic implanted medical device (e.g. pacemaker).
* History of motion sickness within 5 years prior to enrollment will require a tolerability test at baseline.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Adherence rate (acceptability) | 6 weeks
  Adherence will be measured using weekly home practice logs in which participants will record the frequency and duration of their ART-VR exposure. Adherence will be calculated by arm and is defined in arm 1 as using the VR intervention ≥14.4 times (≥432 minutes) over the course of the study. In arm 2, adherence is defined as using the VR intervention ≥19.2 times (≥576 minutes) over the course of the study. The intervention will be considered acceptable if the adherence rate is 80% or more in either arm (or both arms).

SECONDARY OUTCOMES:
Attrition rate (feasibility) | 6 weeks
  Included in the attrition count will be anyone who does not provide response to the Functional Assessment of Cancer Therapy-Cognitive Function (Fact-Cog) questionnaire during week 6 of the study. The intervention will be considered feasible if the attrition rate is 25% or less in either arm (or both arms).
Participant experience assessed using Thematic Analysis | 6 weeks
  During week 6, research staff will record (either via audio or HIPAA-compliant video platform) participant responses to a set of 6 participant experience questions. Responses will be transcribed and reviewed by two study team members. The research team will then connect the codes to try to identify themes for participant experience. Data analysis will be grounded in the theory of Thematic Analysis, which has been proven to be an effective framework for uncovering meaning in qualitative data.
Impact of intervention, measured by Functional Assessment of Cancer Therapy-Cognitive Function (Fact-Cog) questionnaire | At baseline, week 4 and week 6
  Fact-Cog is a 37-item scale with 4 subscales (Perceived Cognitive Impairments, Impact of Perceived Cognitive Impairments on QoL, Comments from Others, Perceived Cognitive Abilities) with a 7-days recall. Effect sizes for the FACT-Cog and subscales will be calculated for each arm from baseline to week 6. Data will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Noel Arring, DNP, PhD, RN, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No